CLINICAL TRIAL: NCT05844501
Title: Inhibition of Small Conductance Calcium-Activated Potassium Current: A New Therapeutic Approach for Atrial Fibrillation
Brief Title: Ondansetron for the Management of Atrial Fibrillation
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: American Heart Association (Other); Purdue University (Other)
Responsible Party: Principal Investigator, James E. Tisdale, Adjunct Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16581; 22TPA964193 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2023-04-13; First posted 2023-05-06 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Atrial Fibrillation
Keywords: Randomized; Placebo-controlled; Ondansetron; Arrhythmias; Atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac | interventions — Ondansetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ondansetron (Experimental): Patients with atrial fibrillation scheduled to undergo AF ablation will receive treatment with ondansetron 8 mg orally twice daily for 28 days (n=40)
  Interventions: Drug: Ondansetron 8mg
- Placebo (Placebo Comparator): Patients with atrial fibrillation scheduled to undergo AF ablation will receive treatment with matching placebo orally twice daily for 28 days (n=40)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ondansetron 8mg — Ondansetron 8 mg orally twice daily for 28 days
  Arms: Ondansetron
Drug: Placebo — Matched placebo orally twice daily for 28 days
  Arms: Placebo

SUMMARY:
"Afib" is a common irregular heartbeat. Afib can cause stroke, blood clots, dementia and death. Medicines used to treat Afib often do not work well and can cause serious side effects. Clinicians need medicines that work better for Afib. Medicines for Afib work by blocking a current in the heart called a potassium current. There is a newer potassium current called IKas that can contribute to Afib. A medicine called ondansetron is used to keep people with cancer from getting sick to their stomach and throwing up. The investigators have found that ondansetron blocks IKas, and the investigators think that this means that ondansetron may work well to treat Afib. So, in this study the investigators want to find out if ondansetron can: 1) Reduce the amount of time that people have Afib, and 2) Slow down the heart rate when people have Afib. The investigators will study 80 people who are scheduled to have an AF ablation. Several weeks prior to undergoing the ablation procedure, these AF patients will be assigned by chance (like flipping a coin) to one of two groups: ondansetron 8 mg by mouth twice daily or a sugar pill (placebo), which they will take for 28 days. The people in the study will not know whether they are receiving ondansetron or placebo. The investigators will find out if ondansetron reduces the percentage of time that people are in Afib. Also, the investigators will find out if ondansetron slows the heart rate while people are having Afib. The investigators will compare the people in the study who take ondansetron with the people in the study who take placebo. This research will help the investigators to find out if ondansetron can be used as a medicine for people who have Afib.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is a common arrhythmia associated with symptoms, stroke, systemic embolism, heart failure, dementia, and mortality. Guideline-recommended strategies for conversion to and maintenance of sinus rhythm (SR) and ventricular rate (VR) control are of limited efficacy and/or are poorly tolerated. There is a critical need for safer, more effective alternatives for AF drug therapy. The apamin-sensitive small-conductance calcium-activated potassium (SK) ion current (IKas) is important for repolarization in the atria and pulmonary vein muscle sleeves. IKas also contributes to sinoatrial and AV node electrophysiology. Therefore, IKas may be a target for rhythm and rate control in AF. Evidence suggests: 1) IKas plays an important role in the mechanism of AF, 2) The antiemetic agent ondansetron at therapeutic concentrations is a potent IKas inhibitor, and 3) Ondansetron is a cardiac-selective IKas inhibitor. Thus, the investigators hypothesize that ondansetron is effective for rhythm and rate control in patients with AF. Specific Aim 1: Determine the efficacy and safety of ondansetron for reducing AF burden. This aim will be achieved via a prospective, randomized, double-blind placebo-controlled study in patients with AF (n=80). Patients with AF scheduled to undergo an elective catheter AF ablation (pulmonary vein isolation) will be randomized in double-blind fashion to receive ondansetron 8 mg twice daily (n=40) or matching placebo (n=40) for 28 days. The study drug/placebo will be initiated several weeks prior to the ablation procedure, and the 28 days of treatment will be complete at least 3 days prior to the ablation. Continuous ECG recording will be performed using 2 consecutive adhesive skin patch ECG monitors, which provide 14-days of continuous recording. The primary outcome measure will be AF burden (percentage of time in AF). Specific Aim 2: Determine the efficacy and safety of ondansetron for VR control in AF. The effect of ondansetron versus placebo on VR control will be assessed. Primary outcome measures will be mean daily heart rates in AF on days 7, 14, 21 and 28 days following initiation of ondansetron/placebo.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18-100 years of age
* ECG-verified AF and/or atrial flutter requiring elective catheter ablation
* Receiving guideline-recommended anticoagulation (if CHA2DS2-VASc score is 0 (men) or 1 (women), anticoagulation can be omitted)

Exclusion Criteria:

* Women of childbearing potential
* Subject reported syncope of unknown origin within the previous 6 months
* Diagnosis of active thyrotoxicosis
* Diagnosis AF from reversible noncardiac causes
* Diagnosis of acutely decompensated heart failure
* Left ventricular ejection fraction less than or equal to 20%

  * New York Heart Association class IV heart failure
  * Diagnosis of severe liver disease (Child-Pugh score greater than or equal to 10)
* Cardiac surgery (preceding 2 months)
* Not receiving anticoagulation due to contraindications (as determined by treating physician and recorded in the medical record)
* Pretreatment QRS > 180 ms, QTc > 450 ms within two weeks of screening visit
* Heart rate < 50 beats per minute in SR
* Diagnosis of hypotension
* Diagnosis of Wolff-Parkinson-White syndrome
* Previous ondansetron hypersensitivity or serotonin syndrome
* Diagnosis of phenylketonuria
* Diagnosis of congenital long QT syndrome
* Concomitant therapy with both beta-blockers and a nondihydropyridine CCB
* History of drug-induced torsades de pointes or QTc prolongation
* Concomitant therapy with QTc-prolonging medications (www.crediblemeds.org), except amiodarone and propafenone
* Concomitant therapy with serotonergic drugs (selective serotonin reuptake inhibitors, serotonin and norepinephrine reuptake inhibitors, monoamine oxidase inhibitors, mirtazapine, lithium, tramadol), apomorphine, phenytoin, carbamazepine, oxcarbazepine, rifampin.
* Left ventricular ejection fraction < 20% and those with NYHA class IV heart failure with reduced ejection fraction (confirmed by diagnosis or echocardiogram within 6 months of enrollment in screening)
* Patients with pre-existing allergies to adhesives
* Patients with neuromuscular stimulators

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Atrial fibrillation burden | Total duration of study (28 days)
  Burden of atrial fibrillation, defined as overall percentage of time in atrial fibrillation.
Ventricular rate control | 7 days after initiation of ondansetron/placebo
  Maximum heart rate while in atrial fibrillation
Ventricular rate control | 14 days after initiation of ondansetron/placebo
  Maximum heart rate while in atrial fibrillation
Ventricular rate control | 21 days after initiation of ondansetron/placebo
  Maximum heart rate while in atrial fibrillation
Ventricular rate control | 28 days after initiation of ondansetron/placebo
  Maximum heart rate while in atrial fibrillation

SECONDARY OUTCOMES:
Proportion of patients in sinus rhythm | 28 days after initiation of ondansetron/placebo
  Proportion of patients in sinus rhythm at 28 days after initiation of ondansetron/placebo
Time to atrial fibrillation recurrence | 28 days after scheduled electrical cardioversion
  Time to atrial fibrillation recurrence after electrical cardioversion
Adverse effects | During the 28 days of treatment with ondansetron or placebo
  Adverse effects associated with ondansetron or placebo

CONTACTS AND LOCATIONS:
Overall Officials: James E Tisdale, PharmD, Principal Investigator — Purdue University
Locations (3):
- United States (3):
  - Indiana Clinical Research Center, Indianapolis, Indiana
  - Indiana University Health Methodist Hospital, Indianapolis, Indiana
  - Purdue University, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR
Time Frame: Data will become available upon publication of study results in clinical trials.gov. Data will be available indefinitely